CLINICAL TRIAL: NCT02023827
Title: Computerized Stage-Matched Intervention for Juvenile Offenders
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pro-Change Behavior Systems (Other)
Collaborators: Iowa Juvenile Court Services (Unknown)
Responsible Party: Principal Investigator, Deborah Levesque, Chief Science Officer, Pro-Change Behavior Systems
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5R44DA024900 (NIH)
Record Dates: First submitted 2013-12-18; First posted 2013-12-30 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Delinquency; Substance Abuse
Keywords: Transtheoretical Model; Stages of change; Computer-tailored intervention; Delinquency; Substance abuse; Juvenile offender; Juvenile justice; Rise Above Your Situation (RAYS) program
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RAYS intervention (Experimental): In addition to standard care, participants receive three monthly online RAYS sessions, each followed by a one-on-one discussion with the probation officer
  Interventions: Behavioral: RAYS Intervention
- Standard care (No Intervention): Participants receive standard care from the probation officer

INTERVENTIONS:
Behavioral: RAYS Intervention — The Rise Above Your Situation program (RAYS) is a multimedia computer-tailored intervention that relies on the Transtheoretical Model of Behavior Change (TTM) and expert system technology to deliver assessments, feedback, printed reports, and helpgiver reports with intervention ideas. Helpgivers (probation officers in this case) use the reports to guide 1/2 hour follow-up discussions to reinforce intervention ideas and provide support.
  Arms: RAYS intervention

SUMMARY:
Juvenile crime imposes enormous costs on victims, on society, and on juvenile offenders themselves. However, research assessing the efficacy of interventions for young offenders show, on average, only small effects on recidivism, substance abuse, and other behavioral outcomes. A major problem with existing interventions is that they tend to neglect individual differences in motivation and readiness to make positive changes. In earlier research, we used an empirically validated model of behavior change, the Transtheoretical Model (TTM, the "stage" model), and expert system technology to develop the Rise Above Your Situation program (RAYS), a prototype of a multimedia computerized tailored intervention designed as an adjunct to traditional juvenile justice programs. The intervention delivers assessments and individualized feedback matched to readiness to stay out of trouble with the law and quit alcohol and drugs. At the end each session the program also generates a helpgiver report that summarizes the youth's feedback and presents concrete, easy-to-implement strategies helpgivers can use to reinforce stage-matched concepts. In the current research, the goals are to complete development of the computerized tailored intervention; develop training and other support materials for helpgivers; and assess the efficacy of the intervention package in a randomized clinical trial involving 700 medium- to high-risk court-involved juveniles aged 13-17 recruited by 54 probation officers randomly assigned to treatment or standard care. Primary outcomes will be criminal recidivism and substance abuse abstinence at 6 and 12 months follow-up.

DETAILED DESCRIPTION:
Fifty-four probation officers employed by the Iowa's Juvenile Court Services agreed to participate in the study and to be randomly assigned to treatment or standard care. A Multiattribute Utility Measurement Approach (Graham, Flay, Johnson, Hansen, & Collins, 1984) was used to ensure that probation officers assigned to the two conditions were approximately equivalent on level of education, years of experience working with juvenile offenders, number of hours of training on the TTM, and confidence using the TTM in their work.

Probation officers were responsible for recruiting moderate- and high-risk youth on probation, and delivering baseline assessment sessions and intervention sessions. However, local project site coordinators were available to provide assistance, as needed.

Computerized follow-up assessments and urine drug testing at 6 and 12 months follow-up are being administered by "trackers" at a time and place that is convenient for the youth. Study protocols include best practices (Scott, 2004) for maximizing retention at follow-up in research involving high-risk populations.

ELIGIBILITY:
Inclusion Criteria:

Juvenile offenders:

* Score in the moderate- to high-risk range on the short-form Iowa Delinquency Assessment
* Age 13 to 17 at the time of recruitment
* Able to understand and read English

Probation officers:

* Employed by Iowa Juvenile Court Services
* Work with moderate- to high-risk youth

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Criminal recidivism based on self-report | 12 months follow-up
  Assessed using the General Crime Scale (GCS) of the Global Appraisal of Individual Needs (GAIN)
Criminal recidivism based on official records | 12 months follow-up
  Data will be provided by the Iowa Division of Criminal and Juvenile Justice Planning (CJJP)
Substance use abstinence based on self-report | 12 months follow-up
  Among youth who screened positive for substance abuse and/or dependence at baseline, assessed using the Substance Frequency Scale (SFS) from the GAIN

SECONDARY OUTCOMES:
Total count of criminal behavior based on self-report | 12 months follow-up
  Assessed using the General Crime Scale (GCS) of the Global Appraisal of Individual Needs (GAIN)
Stage of change for staying out of trouble with the law | 12 months follow-up
  Assessed using a self-report Transtheoretical Model of Behavior Change (TTM) stage of change measure developed by the PI
Emotional distress | 12 months follow-up
  Assessed using the 5-item Internalizing Disorder Screener (IDScr) of the GAIN Short Screener
Substance use frequency | 12 months follow-up
  Among youth who screened positive for substance abuse and/or dependence at baseline, assessed using the Substance Frequency Scale (SFS) from the GAIN
Substance-related problems | 12 months follow-up
  Among youth who screened positive for substance abuse and/or dependence at baseline, assessed using the Substance Problem Scale (SPS) from the GAIN
Stage of change for quitting alcohol and drugs | 12 months follow-up
  Among youth who screened positive for substance abuse and/or dependence at baseline, assessed using a self-report Transtheoretical Model of Behavior Change (TTM) stage of change measure developed by the PI
Abstinence confirmed by urine drug testing | 12 months follow-up
  Among youth who screened positive for substance abuse and/or dependence at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Levesque, Ph.D., Principal Investigator — Pro-Change Behavior Systems, Inc.
Locations (5):
- United States (5):
  - Iowa Juvenile Court Services, District 6, Cedar Rapids, Iowa
  - Iowa Juvenile Court Services, District 7, Davenport, Iowa
  - Iowa Juvenile Court Services, District 5, Des Moines, Iowa
  - Iowa Juvenile Court Services, District 3, Sioux City, Iowa
  - Iowa Juvenile Court Services, District 1, Waterloo, Iowa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levesque DA, Johnson JL, Welch CA, Prochaska JM, Fernandez AC. Computer-Tailored Intervention for Juvenile Offenders. J Soc Work Pract Addict. 2012 Jan 1;12(4):391-411. doi: 10.1080/1533256X.2012.728107. Epub 2012 Nov 8. PMID 23264754